CLINICAL TRIAL: NCT05579821
Title: Evaluation of DPP® Typhoid Assay (Chembio Diagnostic System, Inc) for the Diagnosis of Typhoid From Well Characterized Serum Sample.
Brief Title: Evaluation Study of DPP® Typhoid Assay
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Sponsor
Other Study IDs: FE006C
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Typhoid DPP assay — The index test used in this study diagnose typhoid fever by detecting IgA antibodies against LPS and HlyE antigen in patient's serum.

SUMMARY:
Fever management is a major problem in Low and Middle Income Countries (LMICs) where access to good quality diagnostic test is often unavailable. Fever due to typhoid is similar to other undifferentiated febrile illnesses and typhoid can be mistaken with other vector borne febrile illnesses such as scrub typhus. Currently available diagnostic tests, blood and bone marrow culture, and RDTs have several limitations including a low sensitivity and specificity . Recently, several antigens of Salmonella Typhi useful for serodiagnosis of typhoid has been identified. Salmonella Typhi lipopolysaccharide (LPS) and hemolysin E (HlyE) have been identified as top candidate antigens by several studies to differentiate acute typhoid patients from healthy individuals. DPP® Typhoid Assay is a multiplex rapid test that detects IgA antibodies to LPS and HlyE antigen. It is considered to have high sensitivity and specificity and its results were found to be highly correlated with ELISA results. However, very few studies have been conducted to evaluate this test and limited information about the accuracy of this test is present. Hence, this study will evaluate the sensitivity and specificity of this test in archived serum sample of well characterized blood culture positives and negatives in support of new innovation on typhoid diagnostics.

DETAILED DESCRIPTION:
Typhoid is an acute febrile illness caused by Salmonella enterica serovar Typhi (S. Typhi). Annually, an estimated 11-21 million people become infected with typhoid fever and 128000-161000 people die from the disease . It is commonly transmitted through consumption of contaminated food or water. Low and middle-income countries and areas with poor access to safe water, food and sanitation are at higher risk of infection.

Blood and bone marrow culture is considered as the mainstay for laboratory confirmation of typhoid. However, it is expensive, requires specific laboratory equipment and technical expertise and takes longer time to generate results. Several RDTs and Widal test are available which do not require specialized laboratory and well-trained staff but lack sensitivity and specificity. Several studies have been done for identification of promising antigens that can be used to develop an accurate serodiagnostic assay. S. Typhi lipopolysaccharide (LPS) and hemolysin E (HlyE) have been identified as top candidate antigens by several studies to differentiate acute typhoid patients from healthy individuals. HlyE is a pore-forming toxin that affects bacterial growth within human macrophages and contributes to the cytotoxicity and invasion of epithelial cells.

Dual Path Platform (DPP) Typhoid Assay of Chembio is a point-of-care (POC) immunochromatographic technology which has the capability of measuring IgA response in blood, plasma and serum to both LPS and HlyE. A previous study done on this POC showed promising sensitivity and specificity to diagnose typhoid.Thus, the current study aims to assess the sensitivity and specificity of DPP ® Typhoid Assay using blood culture as the reference point.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria identical to the prior prospective study in AKU (Protocol ref number: FE006)
* Serum stored frozen at AKU as a part of afore mentioned study and cold-chain maintained.

Exclusion Criteria:

* Samples whose reference standard data (Blood culture report) are not available in FIND's OpenClinica database.

Ages: 2 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted at AKU research laboratory using well characterized typhoid positive and typhoid negative serum samples, which were archived for further research purposes from previous trial "Comparative study of commercially available typhoid point of care tests to benchmark current and emerging tools" conducted at AKU in 2020-2021. Precisely, the population is represented by children and adults (age 2-65) who presented with fever of 3-7 days duration.
  All patients from whom these samples were obtained have consented to store their sample at AKU and to use them for research on diagnostic tool for fever management.
  Prospective approval of protocol deviations to recruitment and enrolment criteria, also known as protocol waivers or exemptions, is not permitted.
Sampling Method: Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Point estimates of sensitivity and specificity with 95% confidence interval of DPP Typhoid assay using blood culture as reference standard | October 2022

SECONDARY OUTCOMES:
Estimates of operational characteristics of DPP Typhoid Assay, based on quantitative assessment including invalid rates | Nov 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided